CLINICAL TRIAL: NCT01542216
Title: Evaluation of Nutrition and Metabolism in Breast Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges
Sponsor: University of Waterloo (Other)
Collaborators: Grand River Regional Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17215; 2011-0463 (Other: Tri-Hospital Research Ethics Board)
Record Dates: First submitted 2012-02-20; First posted 2012-03-02 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutritional Status; Exercise; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga and Stretching Group (Placebo Comparator): Patients undergo yoga and stretching exercises
  Interventions: Behavioral: Yoga and Stretching Group
- Nutrition and Exercise Group (Active Comparator): Patients are provided with nutrition, cardiovascular exercise and strength exercise consultations
  Interventions: Behavioral: Nutrition and Exercise Group

INTERVENTIONS:
Behavioral: Nutrition and Exercise Group — Patients randomized to this arm will receive nutrition and exercise consultations. Exercise consultations will home- and institution-based.
  Other Names: Nutrition and Exercise Training
  Arms: Nutrition and Exercise Group
Behavioral: Yoga and Stretching Group — Patients randomized to this arm will receive consultations on yoga and stretching exercises.
  Other Names: Minimal Exercise
  Arms: Yoga and Stretching Group

SUMMARY:
With the increased success in breast cancer therapies, survivors develop unhealthy changes in body composition, such as muscle loss and fat gains, which lead to increased risk of cardiovascular disease and diabetes in survivorship. This study will examine the effects of a nutrition, cardiovascular and strength exercise program compared with a yoga program (representing usual care) on body composition and metabolism in recently diagnosed breast cancer patients. Nutrition and exercise may improve various body composition and metabolic parameters, which may improve quality of life in survivorship, reduce risk of recurrence and reduce the risk of developing cardiovascular disease and diabetes in survivorship.

DETAILED DESCRIPTION:
Despite the increased success of novel anti-neoplastic therapies, breast cancer patients receiving chemotherapy develop unfavourable changes in body composition, including lean tissue loss and fat gains (1,2). These detrimental changes associate with poor quality of life (3,4) and may lead to treatment complications (5,6) during the cancer trajectory. In non-malignant populations, fat gain and muscle loss associate with increased risk of cardiovascular disease and diabetes (7). Cancer survivors who gain fat and lose lean mass are not only predisposed to these diseases but also have an increased risk of cancer recurrence (3). Proper nutrition as well as exercise can independently improve metabolic profiles (i.e. immune function, lipid and glucose metabolism) and overall health outcomes in non-malignant populations (7-9). While exercise has enhanced quality of life in breast cancer patients (4), overall nutritional needs and the metabolic benefits of exercise are unclear in this patient group. Understanding the effects of nutrition and exercise interventions in breast cancer patients will form the basis for future studies and programs that integrate nutrition, exercise, and metabolism to reduce cancer recurrence and other morbidities in survivorship. This study will examine the effects of nutrition and exercise intervention on body composition and metabolism in recently diagnosed breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years old or older
* Recent diagnosis of breast cancer and up to 4 weeks following the first cycle of chemotherapy or up to the first 4 weeks of radiation therapy
* Clinical Stages I-IIIa
* Able to communicate freely in English
* Have sufficient cognitive ability to participate and provide informed consent

Exclusion Criteria:

* Any known diagnosis of cardiovascular disease and thyroid disease that is not currently managed with medication or other therapies
* Any known diagnosis of diabetes or HIV
* Pre-existing injuries or health conditions that prevents the patient's safe participation in exercise
* Any previous diagnosis of cancer within the last 5 years (other than carcinoma in situ)
* Fasting glucose >7.0 mM at baseline of the study
* Pregnant individuals will be excluded from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in glucose parameters from baseline | Baseline, 8 weeks, 16 weeks
  Oral glucose tolerance tests will be performed at each assessment. Changes from baseline will be measured.

SECONDARY OUTCOMES:
Change in lipid profile relative to baseline | Baseline, 8 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marina Mourtzakis, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada